CLINICAL TRIAL: NCT05470491
Title: A Phase I/II Trial of Allogeneic Reduced-Intensity, HLA-Haploidentical Allogeneic Hematopoietic Cell Transplantation Followed by GVHD Prophylaxis With Cyclophosphamide, Bortezomib and Maraviroc for Hematologic Malignancies in People Living With HIV (PLWH)
Brief Title: Trial of Allogeneic Reduced-Intensity, HLA-Haploidentical Allogeneic Hematopoietic Cell Bone Marrow Transplantation Followed by Graft-versus-Host-Disease (GVHD) Prophylaxis With Cyclophosphamide, Bortezomib and Maraviroc for Hematologic Malignancies ...
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10000478; 000478-C
Record Dates: First submitted 2022-07-21; First posted 2022-07-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-26

CONDITIONS: HIV; Hematologic Malignancies
Keywords: Hematopoietic Cell Transplant; HCT; Human Immunodeficiency Virus
MeSH Terms: conditions — Hematologic Neoplasms; Acquired Immunodeficiency Syndrome | interventions — plerixafor; Maraviroc

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/Recipient Arm 1 (Experimental): RIC+alloHCT+GVHD prophylaxis per dose levels 1, 2, and
  Interventions: Drug: RIC; Drug: GVHD prophylaxis; Procedure: allo HCT; Drug: Plerixafor; Drug: Maraviroc
- 2/Recipient Arm 2 (Experimental): RIC+alloHCT+GVHD prophylaxis per RP2D
  Interventions: Drug: RIC; Drug: GVHD prophylaxis; Procedure: allo HCT; Drug: Plerixafor; Drug: Maraviroc
- 3/Donor Arm (No Intervention): Collection of research samples on hematopoietic donors

INTERVENTIONS:
Drug: RIC — e-ATG 40 mg/kg/day IV on days -14 and -13. Prednisone tapering doses given orally daily: -days -14 through -12: 1mg/kg/day -days -11 and -10: 0.75 mg/kg/day -days -9 and -9: 050 mg/kg/day -day -7: 0.25 mg/kg/day Pentostatin 4 mg/m2/day IV on days -11 and -7. Cyclophosphamide 5 mg/kg orally or IV daily on days -11 through -4. Busulfan IV AUC targeted dose of 14.8-23.0 mg*h/L, on days -3 and -2.
  Arms: 1/Recipient Arm 1; 2/Recipient Arm 2
Drug: GVHD prophylaxis — Cyclophosphamide 50 mg/kg IV daily Bortezomib 1.3 mg/m2 IV +6 hours and +72 hours after graft infusion Mesna 50 mg/kg IV concomitant with cyclophosphamide
  Arms: 1/Recipient Arm 1; 2/Recipient Arm 2
Procedure: allo HCT — bone marrow transplant
  Arms: 1/Recipient Arm 1; 2/Recipient Arm 2
Drug: Plerixafor — In phase 1 dose level 3 and phase 2 only: Plerixafor 240 (Micro)g/kg subcutaneously every other day, starting day +1 through day +21
  Arms: 1/Recipient Arm 1; 2/Recipient Arm 2
Drug: Maraviroc — Phase 1 dose level 2: 300 mg orally twice daily starting day-3 through day day+30
  Arms: 1/Recipient Arm 1; 2/Recipient Arm 2

SUMMARY:
Background:

People living with HIV(PLWH) are at a higher risk for cancers that may be curable with a bone marrow transplant. HIV infection itself is no longer a reason to not get a transplant, for patients who otherwise have a standard reason to need transplant.

Objective:

This study is being done to see if a new combination of drugs (cyclophosphamide, maraviroc, and bortezomib) is both safe and effective at protecting against graft-versus-host disease after bone marrow transplant. The study will also test the transplant s impact on your survival and control of your cancer.

Eligibility:

People aged 18 years and older living with HIV and a blood cancer that is eligible for a transplant. Healthy family members aged 12 or older who are half matched to transplant recipients are also needed to donate bone marrow.

Design:

The study will be done in 2 phases. The first phase will be to see if we can safely use a new combination of drugs to prevent GVHD. If the combination is safe in the first phase, the study will proceed to the second phase. In the second phase, we will see if this new combination can better protect against GVHD after transplant.

Participants will be screened. Their diagnoses, organ function and eligibility will be confirmed.

Participants will have a catheter inserted into a vein in their chest or neck. Medications and transfusions will be given through the catheter; blood will be drawn from it.

Participants will be in the hospital for 6 weeks or longer.

They will receive various drugs for 2 weeks to prep their body for the transplant.

The transplant cells will be administered through the catheter.

Participants will continue to receive drug treatments after the transplant.

Blood transfusions may also be needed.

Participants will return 1-2 times per week for follow-up visits for 3 months after discharge.

Participants will have visits 6, 12, 18, 24 months after transplant, then once a year for 5 years.

DETAILED DESCRIPTION:
Background:

* Human Immunodeficiency Virus (HIV) infection should not be considered a barrier to hematopoietic cell transplantation (HCT) in patients who otherwise have a standard indication for HCT.
* The main historical barriers include the risk of opportunistic infections, drug interactions, and lack of donor availability.
* This study addresses these barriers by requiring adequate HIV control with anti-retroviral therapies which do not interact with the transplant medications and by utilizing HLA-haploidentical donors.
* Cellular reservoirs that harbor latent HIV are cells of hematopoietic origin, and thus HCT is a potential cure for HIV if all hematopoietic/immune cells can convert to fully donors without HIV infection of these cells.
* CCR5 receptor and CXCR4 are chemokine co-receptors that enable HIV entry into cells.
* Obtaining a CCR5-delta-32 homozygous donor lacks feasibility for the majority of people living with HIV (PLWH) requiring HCT, particularly those of minority ethnic backgrounds.
* Agents used to prevent graft-versus-host disease (GVHD) include post-transplantation cyclophosphamide (PTCy), maraviroc, and bortezomib

  * PTCy expands the donor pool by allowing HLA-mismatched donor HCT with good engraftment and low rates of GVHD. PTCy typically combined with other agents as adjuncts for GVHD prophylaxis, standardly a calcineurin inhibitor and mycophenolate mofetil
  * Bortezomib has been used in combination with PTCy as GVHD prophylaxis and may additionally inhibit HIV infection of donor cells
  * Maraviroc is used as GVHD prophylaxis, but not previously in combination with PTCy and bortezomib, and is additionally a CCR5 receptor blocker, which may inhibit HIV infection of donor cells. Maraviroc is an HIV medication used in modern ART regimens.
  * This protocol is a step-wise evaluation of a GVHD prophylaxis regimen of PTCy and bortezomib in recipients of HLA-haploidentical grafts among those who are on maraviroc, followed by a de-escalation of maraviroc to serve purely as GVHD prophylaxis
* Plerixafor is used in HCT to promote hematopoietic recovery, akin to the use of G-CSF, and is also a CXCR4 blocker, which may inhibit HIV infection of donor cells

Objective:

* To determine a safe and recommended phase II dose level regimen.
* To determine whether a PTCy-based GVHD prophylaxis regimen including maraviroc and bortezomib can maintain adequate protection against grades III-IV acute GVHD (aGVHD), evaluated at day +100.

Eligibility:

* Transplant recipient: age >= 18 years
* Transplant recipient must be HIV seropositive
* Transplant recipient must have histologically or cytologically confirmed hematologic malignancy with a standard indication for allogeneic HCT, or hematologic malignancy with a standard indication for autologous transplant without access to autologous transplant
* There must be at least one potentially suitable HLA-haploidentical donor.

Design:

* Open-label, single institution, non-randomized, single arm phase II study
* CCR5-delta-32 status will be tested among donor options and homozygous donors will be used, if available
* Conditioning will consist of eATG 40 mg/kg/day IV on days -14 and -13, pentostatin 4 mg/m^2/day IV on days -11 and -7, low-dose cyclophosphamide 5 mg/kg/day orally daily on days -11 through -4; busulfan IV, pharmacokinetically dosed, on days -3 and -2.
* Peripheral blood stem cells are the only graft source allowed for this study.
* GVHD prophylaxis will consist of PTCy 50 mg/kg/day IV on days plus 3 and plus 4, bortezomib 1.3 mg/m^2 IV in 2 doses at 6 and 72 hours after graft infusion for all participants. The phase I will include 2 dose levels of de-escalated maraviroc

  * Dose level 1 - PLWH on a maraviroc-containing ART regimen that starts at least 4 weeks before enrollment and continues at least through day plus100
  * Dose level 2 - PLWH not on a maraviroc-containing ART regimen, treated with maraviroc 300 mg orally twice daily starting day -3 and given through day plus 30 purely for GVHD prophylaxis
* If successful completion of dose level 2, dose level 3 will substitute plerixafor in lieu of G-CSF to the dose level 2 regimen. Plerixafor will be given subcutaneously at 240 microgram/kg every other day, beginning at day plus 1 after transplant through day plus 21, or longer as clinically indicated, such as until ANC recovery.

ELIGIBILITY:
* INCLUSION CRITERIA - RECIPIENT:
* Participants must have a histologically or cytologically confirmed hematologic malignancy with standard indication for allogeneic hematopoietic cell transplantation including, but not limited to, one of the following:

  * Acute myeloid leukemia in morphologic complete remission (<5% blasts in the bone marrow, no detectable abnormal peripheral blasts, and no extramedullary disease)
  * Any secondary and/or treatment related myeloid neoplasm with antecedent history of myeloid neoplasm or previous chemotherapy/radiation
  * B-cell acute lymphoblastic leukemia in first or subsequent complete remission
  * T-cell acute lymphoblastic leukemia in first or subsequent complete remission
  * Myelodysplastic syndrome of intermediate or higher score by the Revised International Prognostic Scoring System (IPSS-R)
  * Primary myelofibrosis of intermediate-2 or higher risk by the Dynamic IPSS-Plus (DIPSS-Plus) or high to very high risk score (5 or higher) calculated with MIPSS70+ Calculator; DIPSS-Plus For Myeloproliferative Neoplasms on the Mutation Enhanced International Prognostic Score System (MIPSS70/MIPSS70+)
  * Chronic myelomonocytic leukemia
  * Chronic myelogenous leukemia resistant to or intolerant of >=3 tyrosine kinase inhibitors or with history of accelerated phase or blast crisis
  * B-cell lymphoma including Hodgkin lymphoma that has relapsed/progressed within 1 year of completion of primary treatment, after autologous transplantation or has progressed through at least 2 lines of therapy
  * Burkitt or lymphoblastic lymphoma: high-risk disease in first remission, progression/relapse after >=1 previous regimen
  * Chronic lymphocytic leukemia with 17p deletion and/or unmutated IgHv or refractory or intolerant of both BTK and PI3K inhibitors
  * Mature T or NK neoplasms as defined in the WHO guidelines of sufficient type and severity for allogeneic HCT based on published clinical practice guidelines
  * T-Prolymphocytic leukemia progressing/relapsing after alemtuzumab and at least one other regimen
  * B-Prolymphocytic leukemia progressing/relapsing after fludarabine and at least one other salvage regimen
  * Hematologic malignancy of dendritic cell or histiocytic cell type
  * Multiple myeloma that relapses after therapy with both a proteasome inhibitor and an immunomodulatory drug (IMiD), relapses after autologous transplantation, or manifests as plasma cell leukemia

In addition to standard indications for HCT: Participant with a hematologic malignancy eligible for consolidation of first remission with autologous transplantation, if autologous transplantation is not accessible to the participant.

* HIV seropositive, with ART regimen that, when stable for >4 weeks, is associated with an HIV viral load <400 copies/mL at screening evaluations. Subsequent changes to avoid/optimize drug interactions with study drugs or essential supportive care drugs may be made to the ART regimen at any time during the eligibility assessment period, as long as the eligibility criteria were met and the regimen change is expected, by the study team and involved consultants/pharmacy, to be similarly effective for HIV control. These changes to the ART regimen are not part of the study. If changes to the ART regimen are made during the eligibility period, HIV viral load will be rechecked at least 1 week after the change but prior to protocol treatment consent.

  * Dose level 1: ART regimen must include maraviroc
  * Dose level 2 and 3: ART regimen must not include maraviroc and there must be no history of maraviroc intolerance or resistance
* Age >= 18 years
* At least one potentially suitable HLA-haploidentical first degree or collateral related donor. Recipients with donor-specific anti-HLA antibodies (DSAs) to all potential donors must have at least one potential donor option where the DSA strength has a mean fluorescence intensity of < 5000 and antibodies are not complement-fixing.
* Karnofsky performance score >=50 percent.
* Adequate organ function defined as possessing all of the following:

  * Cardiac ejection fraction by 2D ECHO of >=40 percent
  * Forced expiratory volume-1 (FEV-1), forced vital capacity (FVC), and diffusing capacity of the lung for carbon monoxide (DLco, adjusted for hemoglobin) all of >=40 percent predicted. If unable to perform pulmonary function tests, there should be no evidence of dyspnea at rest, no requirement for supplemental oxygen, and oxygen saturation >92 percent on room air.
  * Total bilirubin <=3.0 mg/dL (unless due to Gilbert's or hemolysis), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) <= 5x the upper limit of normal, gamma glutamyl transferase (GGT) <= 5x the upper limit of normal
* Estimated serum creatinine clearance of >=50 mL/min/1.73m2 calculated using eGFR in the clinical lab
* Ability of participant to understand and the willingness to sign a written informed consent document.
* Individuals of childbearing potential and those that can father children must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for at least one-year post-allo HCT.

EXCLUSION CRITERIA - RECIPIENT:

* Participants who are receiving any other investigational agents that cannot be discontinued/completed at least 2 weeks prior to the date of beginning conditioning.
* Poorly controlled malignant indication for transplantation, defined as:

  * Leukemia not having achieved morphologic remission (i.e. bone marrow blasts >5 percent or active extramedullary disease)
  * Lymphoma not having demonstrated some degree of treatment sensitivity (chemosensitivity, radiosensitivity) by clinical and/or radiologic assessment
  * Multiple myeloma not in complete remission, as determined by negative immunofixation in serum and urine and disappearance of any soft tissue plasmacytomas and <= 5 percent plasma cells in the bone marrow.
* Uncontrolled intercurrent illness that in the opinion of the PI would make it unsafe to proceed with transplantation.
* Study team is unable to identify an adequate antiretroviral regimen to adequately suppress the HIV viral load <400 copies/mL that is compatible with study drugs
* Pregnancy
* For lactating potential participants: unwilling to discontinue lactation prior to the start of study treatment on day -14.
* Prohibitive allergy to a study drug or to compounds of similar chemical or biologic composition of the agents (eATG, steroids, cyclophosphamide, busulfan, pentostatin, maraviroc, bortezomib, plerixafor (dose level 3 only)) used in the study.
* Lack of central access potential sufficient for transplant
* Active psychiatric disorder which is deemed by the PI to have significant risk of compromising compliance with the transplant protocol and/or antiretroviral therapy
* Grade 3-4 motor or sensory neuropathy per CTCAE version 5.0

INCLUSION CRITERIA - RELATED DONOR:

* Related donor (age >=12) deemed suitable and eligible, and willing to donate, per clinical evaluations, who are additionally willing to donate blood and/or PBSC graft aliquotfor research. Related donors will be evaluated in accordance with existing institutional Standard Policies and Procedures for determination of eligibility and suitability for clinical donation.
* Ability of participant or parent/legal guardian to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA - RELATED DONOR:

-Failure to qualify per institutional Standard Policies

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 265 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
In phase II, avoidance rate of grade III-IV acute GVHD at day +100 | day +100 post HCT
  Proportion of evaluable recipients who experience grade III-IV acute GVHD at day +100 will be reported along with 80% and 95% two-sided confidence interval
Determine a safe and recommended phase II dose level regimen | day +100 post HCT
  Number and type of toxicities noted for participants who are evaluable

SECONDARY OUTCOMES:
Cumulative incidence of primary and secondary graft failure | day +100 and 1 year post HCT
  Cumulative incidence of primary and secondary graft failure based on chimerism at day +100 and 1 year post transplant
Cumulative incidence of hematopoietic recovery | day +100
  cumulative incidence of hematopoietic recovery will be based on platelet recover at day +100
Overall Survival | 1, 2, 3, 4, and 5 years post HCT
  Time from transplant to death of any cause and will be determined using the Kaplan-Meier method
Cumulative incidence of relapse | 1, 3, and 5 years post HCT
  Cumulative incidence rates will be estimated based on disease-risk index.
GVHD-free, relapse free survival (GRFS) | 1, 3, and 5 years post HCT
  Time from transplant to death from any cause of other event and will be determined using the Kaplan-Meier method
Cumulative incidence of acute GVHD | Day +180 and 1 year post HCT
  Evaluation by all grades, grade II-IV, and grade III-IV
Cumulative incidence of chronic GVHD | 1 and 2 years post HCT
  Evaluation by severity of mild, moderate, and severe
Progression Free Survival (PFS) | 1, 3, and 5 years post HCT
  Time from transplant to disease progression and will be determined using the Kaplan-Meier method
Cumulative incidence of transplant-related mortality (TRM) | day +100, 1 year, and 2 years post HCT
  cumulative incidence of transplant related mortality will be estimated

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa A Hyder, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGAP
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as the database is active
Access Criteria: Clinical data will be made available via subscription to BTRIS and with permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000478-C.html